CLINICAL TRIAL: NCT00712179
Title: Developing Evidence-based Parameter Selection for Locomotor Training
Brief Title: Understanding Different Parameters in Locomotor Training (a Type of Walking Training) for Person After a Stroke
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: A6365-R
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Results first posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Stroke
Keywords: Stroke; walking; Treadmill; body weight support system
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke Survivors: Subjects walked with or with therapists' assistance at different speeds and different amounts of body weight support across conditions.

SUMMARY:
This is a research study to understand how people who have experienced a stroke walk in order to develop better and more effective types of therapy. Data collected from people who have experienced a stroke and healthy individuals will be used to compare a neurologically healthy person to someone, which has sustained an injury.

DETAILED DESCRIPTION:
The first day will be a chance for the participants to become familiar with the body weight support (BWS) system and walking at different speeds. This first day will last about 2 hours and will consistent of fifteen total minutes of locomotor training utilizing manual trainers. This means trainers will move the participants'' body into a more normal walking pattern. The participants will be given a chance to rest between bouts; however, the participants may also rest at any point.

First, the participants will walk for five minutes at normal comfortable speed with 15% of the body weight supported through an overhead system. This will be followed by walking at speeds faster and slower than the participants' comfortable speed. After these initial bouts of stepping, will be the training bouts. Training will be conducted with 30% of the body weight supported and at speeds considered normal for adults. Trainers will assist the trunk and with each leg, and will assist with initiation of steps and leg positioning, maintenance of an upright trunk, pelvic rotation, and weight shift. Training will consist of three bouts of five minutes of stepping for a total duration of 15 minutes of stepping. Vital signs, heart rate and blood pressure, will be monitored after each 5-minute bout. If the participants wear an Ankle Foot Orthosis (AFO), the participants will be asked to walk without it, but the investigators will provide the participants with an Aircast, which supports the ankle and prevents it from rolling side to side, but allows the foot to move freely up and down ,

Data will be collected on the second day. This will take approximately five hours. During this time the participants will be asked to walk on the ground and on a treadmill. For the overground portion, the participants will walk across a 14-foot level, pressure-sensitive walkway at the participants' own speed and then as fast as the participants' can safely. This walkway measures the speed of walking and the size of steps. The participants can use any assistive device that the participants' typically use. A physical therapist or trained assistant will walk beside as the participants walk across the walkway. The participants will be asked to walk several times across the walkway at the two speeds while recordings are made from the participants' muscles and are videotaped.

The participants will also be asked to walk on a treadmill. The participants will be permitted to practice treadmill walking until the participants' feel comfortable. Once the participants feel comfortable the investigators will ask the participants to walk a couple different ways. The order will be random, and the speeds will be determined from the first visit. The participants will be asked to walk some with Body Weight Support and some without. The investigators will ask the participants to walk at the participants' comfortable speed and then as fast as the participants' can safely walk. The participants will also walk at these same speeds and percentage of body weight support while trainers help the participants step in a way as close to normal.

The participants will be able to rest at any point and for as long as they wish, however, after each trial the participants will be required to rest at least 2 minutes.

During all treadmill walking, the participants will wear a harness attached to a mobile device attached to the ceiling. This device is for safety to prevent a fall and it can catch the participants should they lose balance or stumble. It will also be used to provide body weight support for some of the walking trials. If the participants use braces and/or assistive devices, the participants will be asked to do some walking with and without them, according to the participants' comfort and safety. A therapist will walk with the participants to provide any physical assistance that may be needed.

For the walking testing, the investigators may need to shave small areas of the participants' legs to attach small sensors to the skin to measure the electrical activity of the leg muscles. The investigators will also attach reflective markers or small angle measurement devices to the skin over the participants' hips and several locations on the legs. The investigators will film the participants' movements with video cameras.

ELIGIBILITY:
Inclusion Criteria:

* adults at least 18 years old;
* able to provide informed consent;
* able to follow three-step motor command;
* have a single unilateral stroke;
* medically stable (i.e. asymptomatic for bladder infection, decubiti, osteoporosis, cardiopulmonary disease, pain, or other significant medical complications that would prohibit or interfere with walking;
* able to stand with assistance and/or ambulate 15 meters with or without an assistive device or brace and no greater than standby physical assistance.

Exclusion Criteria:

* weight > 300 pounds due to limitations in body weight support systems;
* body size which is incompatible with harnesses;
* pregnancy;
* presence of significant musculoskeletal problems that limit hip and knee extension or ankle plantarflexion to neutral;
* self selected walking speed below 0.3 m/s; and
* history of congestive cardiac failure, unstable angina, or peripheral vascular disease.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Controls and persons who have sustained a stroke
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve A. Kautz, PhD MS BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Srivastava S, Patten C, Kautz SA. Altered muscle activation patterns (AMAP): an analytical tool to compare muscle activity patterns of hemiparetic gait with a normative profile. J Neuroeng Rehabil. 2019 Jan 31;16(1):21. doi: 10.1186/s12984-019-0487-y. PMID 30704483

RESULTS

PARTICIPANT FLOW:
Groups:
- Stroke Survivors: Stroke survivors walked with varying speeds, amount of body weight support or therapist assistance
Period: Overall Study
Arm/Group | Stroke Survivors
Started | 49
Completed | 37 (Data from 4 subjects was excluded due to noise in recorded EMG signal, so 33 subjects were analysed.)
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- Stroke Survivors: Cross-sectional study with a single group of stroke survivors
Arm/Group | Stroke Survivors
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 49
Baseline walking speed [Mean (Standard Deviation); unit: meters per second] | 0.59 (0.23)

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic
Description: The electromyographic (EMG) gait pattern of stroke survivors was compared with "normal" pattern using z-scores.
Time Frame: During sessions- 1 day measurement
Population: Individuals with chronic stroke.
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Stroke Survivors
Number analyzed (Participants) | 33
Z-score
  Walking at different speeds with 15% BWS | 1.57 (0.058)
  Walking at self-selected speed at 0%, 15%, 30% BWS | 1.57 (0.072)
  Walking at different speeds with 30% BWS | 1.55 (0.075)
  Fastest comfortable speed with different BWS | 1.56 (0.073)
  Modified non-paretic leg loading and movement | 1.64 (0.079)
  Modified paretic leg loading and movement | 1.38 (0.061)
Statistical Analysis 1: Comparison: Stroke Survivors; Null Hypothesis: Walking at different speeds with 15% body weight support will have no effect on EMG pattern; Test type: Superiority or Other; p = 0.981, Mixed Models Analysis
Statistical Analysis 2: Comparison: Stroke Survivors; Null Hypothesis: Walking at self selected speed at 0%, 15% and 30% of body weight support will have no effect on EMG pattern; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis
Statistical Analysis 3: Comparison: Stroke Survivors; Null Hypothesis: Walking at different speeds with 30% body weight support will have no effect on EMG pattern; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis
Statistical Analysis 4: Comparison: Stroke Survivors; Null Hypothesis: Walking at fastest comfortable speeds with different amount of body weight supports will not affect the EMG pattern; Test type: Superiority or Other; p = 0.073, Mixed Models Analysis
Statistical Analysis 5: Comparison: Stroke Survivors; Null Hypothesis: Modification of non-paretic leg loading and movement by the therapist will have no effect on EMG pattern of paretic leg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 6: Comparison: Stroke Survivors; Null Hypothesis: Modification of paretic leg loading and movement by the therapist will have significant effect on EMG pattern of non-paretic leg; Test type: Superiority or Other; p = 0.94, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Stroke Survivors
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No